CLINICAL TRIAL: NCT03235661
Title: Bi-level Positive Airway Pressure for Respiratory Distress Syndrome in Twins:A Randomized Controlled Trials
Brief Title: Bi-level Positive Airway Pressure for Respiratory Distress Syndrome in Twins Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ma Juan, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: twins with BiPAP
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: nCPAP; BiPAP; Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: BiPAP and nCPAP are used as primary mode of ventilation in preterm twins infants with RDS
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BiPAP (Experimental): BiPAP as a primary mode of ventilation in one of the preterm infants with respiratory distress syndrome
  Interventions: Device: BiPAP
- nCPAP (Active Comparator): nCPAP is used as a primary mode of ventilation in another of the preterm infants with respiratory distress syndrome
  Interventions: Device: nCPAP

INTERVENTIONS:
Device: BiPAP — BiPAP is used as a primary mode of ventilation in one of the preterm infants with respiratory distress syndrome
  Arms: BiPAP
Device: nCPAP — nCPAP is used as a primary mode of ventilation in another of the preterm infants with respiratory distress syndrome
  Arms: nCPAP

SUMMARY:
The investigators compared advantages and disadvantages of two forms of noninvasive respiratory support -bi-level positive airway pressure(BiPAP) or nasal continuous positive airway pressure (nCPAP) -as a primary mode of ventilation in preterm twins infants with respiratory distress syndrome

DETAILED DESCRIPTION:
Invasive ventilation is related to development of adverse pulmonary and nonpulmonary outcomes in ventilated infants. Various modes of noninvasive respiratory support are being increasingly used to minimize the incidence of bronchopulmonary dysplasia (BPD). The aim of this trial to compare the effects of bi-level positive airway pressure(BiPAP) and nasal continuous positive airway pressure (NCPAP) in preterm twins infants as the primary mode.

ELIGIBILITY:
Inclusion Criteria:

* 1. Gestational age (GA) is from 26 to 37 weeks;
* 2. Diagnosis of respiratory distress syndrome. The diagnosis of respiratory distress syndrome will be based on clinical manifestations (tachypnea, nasal flaring and or grunting) and chest X-ray findings;
* 3. Respiratory distress syndrome Silverman score >5;
* 4. Informed parental consent has been obtained.

Exclusion Criteria:

* 1. Severe respiratory distress syndrome requiring early intubation according to the American Academy of Pediatrics guidelines for neonatal resuscitation;
* 2. Major congenital malformations or complex congenital heart disease;
* 3. Group B hemolytic streptococcus pneumonia, septicemia, pneumothorax, pulmonary hemorrhage;
* 4. Cardiopulmonary arrest needing prolonged resuscitation;
* 5. transferred out of the neonatal intensive care unit without treatment.

Ages: 5 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
intubation rate | within 7 days
  the baby was intubated

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD,MD, Study Director — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Department of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided